CLINICAL TRIAL: NCT02191033
Title: Text Messaging to Augment Physician Brief Advice for Smoking Cessation in College Health Clinics
Brief Title: Text Messaging for Smoking Cessation in College Health Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Southern Connecticut State University (Unknown); University of New Haven (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1404013813
Record Dates: First submitted 2014-07-08; First posted 2014-07-15 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Cigarette Smoking
Keywords: cigarette smoking; tobacco use cessation products
MeSH Terms: conditions — Cigarette Smoking | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Text messaging (Experimental): Smoking counseling, nicotine patch, text messaging
  Interventions: Behavioral: Smoking counseling; Behavioral: Text messaging; Drug: Nicotine patch
- Standard of care (Active Comparator): Smoking counseling, nicotine patch
  Interventions: Behavioral: Smoking counseling; Drug: Nicotine patch

INTERVENTIONS:
Behavioral: Smoking counseling
Behavioral: Text messaging
  Arms: Text messaging
Drug: Nicotine patch

SUMMARY:
This study is a randomized-controlled clinical trial which evaluates the efficacy of physician brief advice, nicotine replacement therapy and a 6-week course of text messaging in promoting cigarette smoking in smokers enrolled in college.

The primary hypothesis is that smokers receiving physician brief advice, nicotine replacement therapy, and text messaging will have higher quit rates that smokers receiving physician brief advice and nicotine replacement therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 through 24 years
* Enrolled as a full/part time college student
* A current smoker (Have smoked more than 100 cigarettes in their lifetime and now smoke every day or some days)
* English-speaking
* Interested in quitting
* Have a cell phone for personal use with an unlimited text messaging plan.

Exclusion Criteria:

* History of hypersensitivity/allergy to nicotine patch;
* Serious arrhythmias - History of heart disease (myocardial infarction, severe chest pain, or coronary artery disease)
* Current pregnancy/breastfeeding/plan for pregnancy

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepa R Camenga, MD, Principal Investigator — Yale University
Locations (1):
- Southern Connecticut State University, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment open from January 2015 to May 2016. Recruited from local college campuses.
Groups:
- Text Messaging: Smoking counseling, nicotine patch, text messaging
  Smoking counseling
  Nicotine patch
  Text messaging
- Standard of Care: Smoking counseling, nicotine patch
  Smoking counseling
  Nicotine patch
Period: Overall Study
Arm/Group | Text Messaging | Standard of Care
Started | 20 | 20
Completed | 18 | 19
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Text Messaging: Smoking counseling, nicotine patch, text messaging
  Smoking counseling
  Text messaging
  Nicotine patch
- Total: Total of all reporting groups
Arm/Group | Text Messaging | Standard of Care | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.9 (1.7) | 20.5 (1.5) | 20.2 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 7 | 11 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 17 | 19 | 36
  Race: Black | 2 | 0 | 2
  Race: Asian | 1 | 0 | 1
  Race: American Indian/Alaskan Native | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Study Enrollment- Number of Participants Who Join the Study
Description: We will report the number of persons who join the study.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Text Messaging | Standard of Care
Number analyzed (Participants) | 20 | 20
Participants | 20 | 20

2. Primary Outcome: Study Retention- Number of Participants Who Attend the 6- and 12-week Follow up Visits.
Description: We will determine the number of enrolled participants who follow up at the 6- and 12- week follow up visit.
Time Frame: 6- and 12- weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Text Messaging | Standard of Care
Number analyzed (Participants) | 20 | 20
Participants
  6-week retention | 19 | 20
  12-week retention | 19 | 18

3. Secondary Outcome: Smoking Abstinence
Description: biochemically confirmed point prevalence of self reported past 7-day abstinence
Time Frame: 6- and 12- weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Text Messaging | Standard of Care
Number analyzed (Participants) | 20 | 20
Participants
  6-week | 3 | 5
  12-week | 1 | 1

ADVERSE EVENTS:
Time Frame: From January 2015 through August 2016
Arm/Group | Text Messaging | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
This is a pilot and feasibility study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No